CLINICAL TRIAL: NCT02631382
Title: Wet Cupping (AlHijamah); Double Versus Single Cupping Technique in Chronic Low Back Pain Patients: Randomized Comparative Clinical Trial, Pilot Study Saudi Arabia, 2015
Brief Title: Wet Cupping (AlHijamah); Double Versus Single Cupping Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Alternative Medicine, Saudi Arabia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NCCAM - TRIAL - CUPPING2
Record Dates: First submitted 2015-12-06; First posted 2015-12-16 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2015-12

CONDITIONS: Low Back Pain
Keywords: wet cupping Saudi Arabia
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wet cupping : double cupping (Experimental): wet cupping: (traditional cupping technique): cupping (suction) - Scarification - cupping (suction)
  Interventions: Procedure: wet cupping
- wet cupping: single cupping (Experimental): wet cupping:(Asian cupping): Puncture by needles then cupping (suction):
  Interventions: Procedure: wet cupping

INTERVENTIONS:
Procedure: wet cupping — In double cupping (traditional technique): Cupping (suction) then scarification then cupping (suction).
  In single cupping (Asian): puncture using auto lancet then cupping (suction). In both techniques 4 out of 6 acupoints (BL23, BL24, BL25 bilateral) will be selected.
  Other Names: Hijamah; wet cupping device

SUMMARY:
Randomized clinical trial to compare the effectiveness and safety of double (traditional) versus single (Asian) cupping techniques in chronic low back pain.

DETAILED DESCRIPTION:
Chronic Low Back Pain is a very common pain disorder in the primary care. As in many chronic pain conditions, patients are usually asking for alternative options, especially local traditional and therapies including wet cupping, to replace the long-term use of painkillers. The majority of the wet cupping trials conducted abroad used different techniques, which is different from our local traditional wet cupping technique. This study can identify the technique that is more efficacious in reducing pain, prolonging the pain relieve period, and decrease patient dependence on painkillers in chronic low back pain.The aim of this study is to compare the effectiveness and safety of double (traditional) versus single (Asian) cupping techniques in chronic low back pain. This a randomized comparative effectiveness pilot clinical trial. After taking written informed consent, patient with chronic low back pain will be randomized into two groups, one group to receive wet cupping therapy with the Traditional double technique, the other group to receive it with the Asian single technique. Numeric Rating Scale, Present Pain Intensity and Oswestry Disability Questionnaire will be used to measure the outcome before and after the intervention, one week after the intervention, then two weeks after. Wilcoxon rank sum test for the continuous dependent data analysis and the analysis of covariance ANCOVA, to compare both groups mean scores will be used. The outcome baseline for each score will be used as the covariate. Chi square or Fisher's exact test will be used to compare categorical data with Minimal Clinical Improvement Difference within and between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Age equal or more than 18 years up to 60 years
* Chronic low back pain (at least the duration ≥ 3 months)
* Not on anti-inflammatory or pain killers for the last 15 days.

Exclusion Criteria:

* Patients received wet-cupping therapy before in the last three months
* Patients who have low back pain due to specific and known etiological causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome, and cauda equinal syndrome)
* Patients who are inappropriate to the wet cupping treatment (AIDS, Hepatitis, Tuberculosis, Syphilis. The referring physicians will be advised to exclude those patients)
* Patients currently receiving any anticoagulant, antiplatelet medications
* Anemia, thrombocytopenia, Coagulopathy or Hemorrhagic disease like hemophilia
* Had undergone a surgery, or had bleeding injury, or had blood donation
* Uncontrolled hypertension, Ischemic heart disease, previous transient ischemic attack or stroke
* Diabetes, known renal and / or hepatic diseases
* Patients who are in pregnancy or have plan to conception
* Previously or currently drug addicts
* Any other severe disease or disabling medical condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pain Numeric rating scale (NRS) before and after intervention | 14 DAYS
  numeric pain scale to be measured before intervention then two weeks after

SECONDARY OUTCOMES:
pain: McGill, Persistent Pain Intensity (PPI) | 14 days
  before intervention and two weeks later
functioning (Disability) using the Oswestry Disability Questionnaire (ODQ) | 14 days
  functionality will be measured using the questionnaire and compared two weeks after intervention
the Safety of the two wet cupping techniques, by collecting safety data after two weeks of the intervention | up to 14 days
  using the WHO guidelines for classification of adverse events

OTHER OUTCOMES:
Patient satisfaction using the Integrative Medicine Patient Satisfaction Scale (IMPSS) | up to 14 days
  5 grade scales will be compared to a five grade scales of expectation measured before intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sulaiman AlEidi, MBBS, Principal Investigator — NCCAM , MOH, Riyadh, Saudi Arabia; Mohamed Khalil, MD, Study Chair — NCCAM.MOH; Ashry Gad Mohamed, MD, Study Chair — King Saud University
Locations (2):
- Saudi Arabia (2):
  - King Fahad Hospital, Jeddah, Jeddah
  - King Fahad Hospital, Madinah, Madinah

IPD SHARING:
Plan to Share IPD: Undecided